CLINICAL TRIAL: NCT02105558
Title: Outcomes of Epidural Versus Combined Spinal and Epidural (CSE) Anesthetic Technique on the Success of Trial of Labor After Cesarean (TOLAC): A Pilot Study
Brief Title: Outcomes of Neuraxial Anesthetic Technique on the Trial of Labor After Cesarean (TOLAC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jennifer Lynne Erian, Resident, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-14-0023
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Labor Pain; Complications; Cesarean Section; Pregnancy
Keywords: trial of labor after cesarean; vaginal birth after cesarean; epidural vs combined spinal epidural
MeSH Terms: conditions — Labor Pain | interventions — Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epidural anesthesia (Experimental): Trial of labor after cesarean with an epidural for anesthesia: Epidurals will be placed in a sterile fashion using a 17g Tuohy needle to locate the epidural space via loss-of-resistance to saline at the lumbar vertebral level. 3 ml of 1.5% lidocaine with 5ug/ml of epinephrine will then be used for test dose to exclude intrathecal or intravenous placement of the catheter. Epidural solution composed of 5ml of 0.2% ropivacaine and another 5 ml of 0.2% ropivacaine will then be administered.
  Interventions: Drug: Epidural anesthesia
- Combined spinal and epidural anesthesia (Experimental): Trial of labor after cesarean with a combined spinal and epidural (CSE) for anesthesia: the epidural space will be located with a 17g Tuohy needle and dural puncture performed with 25g Pencan needle via needle-through-needle technique. Spinal injection of 2ml 0.2% ropivacaine will then be performed and spinal needle removed. An epidural catheter will then be placed and test dose performed with 3 ml of 1.5% lidocaine with 5ug/ml of epinephrine. Maintenance dose will be via an epidural pump using 0.2% ropivacaine at a rate of 12 ml/hr.
  Interventions: Drug: Combined spinal and epidural anesthesia

INTERVENTIONS:
Drug: Epidural anesthesia — ￼An epidural involves injecting pain-blocking medication into a space between the vertebrae and the spinal fluid; it usually takes about 15 minutes to work.
  Epidurals will be placed in a sterile fashion using a 17g Tuohy needle to locate the epidural space via loss-of-resistance to saline at the lumbar vertebral level. 3 ml of 1.5% lidocaine with 5ug/ml of epinephrine will then be used for test dose to exclude intrathecal or intravenous placement of the catheter. Epidural solution composed of 5ml of 0.2% ropivacaine and another 5 ml of 0.2% ropivacaine will then be administered.
  Arms: Epidural anesthesia
Drug: Combined spinal and epidural anesthesia — A spinal is an injection directly into the spinal fluid; it is given in addition to the epidural technique and takes effect in five minutes.
  The epidural space will be located with a 17g Tuohy needle and dural puncture performed with 25g Pencan needle via needle-through-needle technique. Spinal injection of 2ml 0.2% ropivacaine will then be performed and spinal needle removed. An epidural catheter will then be placed and test dose performed with 3 ml of 1.5% lidocaine with 5ug/ml of epinephrine. Maintenance dose will be via an epidural pump using 0.2% ropivacaine at a rate of 12 ml/hr.
  Arms: Combined spinal and epidural anesthesia

SUMMARY:
To compare the effects of epidural versus combined spinal and epidural (CSE) anesthesia on the success of Trial of Labor After Cesarean (TOLAC).

DETAILED DESCRIPTION:
Though it has been said, "once a cesarean, always a cesarean," the current medical stance has changed and now encourages vaginal birth after cesaren (VBAC) in a select population of patients. VBAC has several advantages over a repeat cesarean including decreased recovery period, decreased risk of infection, avoidance of major abdominal surgery, and lessened blood loss. Predictors for success of VBAC include previous spontaneous vaginal birth, singleton pregnancy, and previous low transverse scar for C-section delivery. TOLAC is a reasonable option for select pregnant women and is associated with a 74% likelihood of VBAC. Risk factors for failure of VBAC include labor dystocia, advanced maternal age, maternal obesity, fetal macrosomia, gestational age (GA) >40 weeks, short inter pregnancy interval, and preeclampsia.

While success of VBAC is associated with fewer complications, failure of VBAC may be associated with increased complications. A major concern for VBAC is the possibility for uterine rupture, which may result in hysterectomy and intrapartum fetal hypoxia/death. According to the American College of Obstetricians and Gynecologists (ACOG) guidelines, effective regional analgesia should not be expected to mask the signs and symptoms of uterine rupture, particularly because the most common sign of rupture is fetal heart tracing abnormalities. Adequate pain relief achieved with either CSE or epidurals may even encourage more women to opt for VBAC. The decision to proceed with TOLAC should occur only after appropriate discussion of the risks and benefits has occurred between the patient and her obstetrician and as long as no other contraindications exist. The final decision should be left up to the patient. There is no reliable way to predict risk of uterine rupture, but it may be associated with classical and low vertical uterine scars, induction of labor, and increased number of prior cesarean deliveries and risk may be decreased by previous vaginal birth. Other aspects of VBAC versus repeat cesarean pertaining to the fetus to consider include respiratory function, mother-infant contact, and initiation of breastfeeding, which may be delayed in cesarean deliveries.

There is very little research concerning the effects of CSEs and epidurals on women undergoing TOLAC.There have been multiple studies comparing CSE and epidurals on nulliparous and multiparous women, but none have been done specifically on patients undergoing TOLAC. According to the American Society of Anesthesiologists (ASA) practice guidelines for obstetric anesthesia "nonrandomized comparative studies suggest that epidural analgesia may be used in a trial of labor for previous cesarean delivery patients without adversely affecting the incidence of vaginal delivery. Randomized comparison of epidural versus other anesthetic techniques were not found." They agree that neuraxial techniques improve the likelihood of vaginal delivery for patients attempting VBAC and suggest neuraxial catheter be placed in event of operative delivery. Because no study to date has compared CSEs and epidurals and their effects on the success of VBAC, this study aims to further investigate this arena.

ELIGIBILITY:
Inclusion Criteria:

* all patients meeting ACOG guidelines for TOLAC
* at least one previous elective cesarean delivery
* <40 weeks gestational age (GA)
* vertex singleton pregnancy with use of continuous fetal monitoring

Exclusion Criteria:

* Patient refusal of regional anesthetic or with contraindication for regional anesthesia
* BMI >40
* associated comorbidities such as gestational diabetes, preeclampsia, abnormal placentation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-04; Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Opal Raj, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Lyndon B. Johnson Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 were enrolled, but only 43 started. Of the 3 who did not start: 1 gave birth before the block placement; 2 were disenrolled, but the reason was not recorded.
Groups:
- Epidural Anesthesia: ￼An epidural involves injecting pain-blocking medication into a space between the vertebrae and the spinal fluid; it usually takes about 15 minutes to work.Epidurals will be placed in a sterile fashion using a 17g Tuohy needle to locate the epidural space via loss-of-resistance to saline at the lumbar vertebral level. 3 ml of 1.5% lidocaine with 5ug/ml of epinephrine will then be used for test dose to exclude intrathecal or intravenous placement of the catheter. Epidural solution composed of 5ml of 0.2% ropivacaine and another 5 ml of 0.2% ropivacaine will then be administered.
- Combined Spinal and Epidural (CSE) Anesthesia: A spinal is an injection directly into the spinal fluid; it is given in addition to the epidural technique and takes effect in five minutes.
  The epidural space will be located with a 17g Tuohy needle and dural puncture performed with 25g Pencan needle via needle-through-needle technique. Spinal injection of 2ml 0.2% ropivacaine will then be performed and spinal needle removed. An epidural catheter will then be placed and test dose performed with 3 ml of 1.5% lidocaine with 5ug/ml of epinephrine. Maintenance dose will be via an epidural pump using 0.2% ropivacaine at a rate of 12 ml/hr.
Period: Overall Study
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Started | 15 | 28
Completed | 15 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia | Total
Number analyzed (Participants) | 15 | 28 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (6.1) | 27.6 (5.9) | 27.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 28 | 43
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 27 | 40
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 28 | 43
Reason for Previous Cesarean [Count of Participants; unit: Participants]
  Breech | 5 | 4 | 9
  Hydrocephalus | 1 | 0 | 1
  Non-reassuring fetal heart tone | 0 | 4 | 4
  Preterm premature rupture of the membranes (PPROM) | 1 | 0 | 1
  Macrosomia | 0 | 2 | 2
  Failure to progress | 3 | 5 | 8
  Oligohydramnios | 0 | 2 | 2
  Congenital fetal heart anomaly | 0 | 1 | 1
  Pre-eclampsia | 0 | 1 | 1
  Scoliosis, nuchal cord | 1 | 0 | 1
  Chorioamnionitis | 0 | 1 | 1
  Macrosomia, breech | 0 | 1 | 1
  Placenta previa | 0 | 1 | 1
  Fetal bradycardia | 0 | 2 | 2
  Low amniotic fluid | 0 | 1 | 1
  Fetal distress | 1 | 1 | 2
  Arrest of labor | 0 | 1 | 1
  Nuchal cord | 0 | 1 | 1
  Malpresentation | 1 | 0 | 1
  Failed induction | 1 | 0 | 1
  Gastrochisis | 1 | 0 | 1
Number of pregnancies [Mean (Standard Deviation); unit: number of pregnancies] | 3.3 (1.6) | 3.0 (0.9) | 3.1 (1.3)
Estimated fetal weight [Mean (Standard Deviation); unit: grams] | 3484 (279) | 3264 (400) | 3341 (374)
Actual fetal weight [Mean (Standard Deviation); unit: grams] — Population: Actual birth weight was not recorded for one in the Epidural anesthesia group.
  grams
    number analyzed (Participants) | 14 | 28 | 42
    (all) | 3453 (445) | 3292 (369) | 3346 (398)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vaginal Birth After Cesarean (VBAC)
Time Frame: at the time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 15 | 28
Participants | 12 | 22

2. Secondary Outcome: Success of Analgesia as Indicated by Pain Score Assessed by Visual Analogue Scale (VAS)
Description: Pain score was assessed by a visual analogue scale (VAS) with a scale of 1 to 10, with higher scores indicating a higher level of pain. Pain scores less than 3 are considered to indicate successful analgesia.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 15 | 28
units on a scale | 7.53 (2.64) | 8.20 (1.89)

3. Secondary Outcome: Success of Analgesia as Indicated by Pain Score Assessed by Visual Analogue Scale (VAS)
Description: as for outcome 2
Time Frame: 15 minutes after regional anesthesia
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 15 | 28
units on a scale | 2.80 (2.08) | 2.13 (2.30)

4. Secondary Outcome: Success of Analgesia as Indicated by Pain Score Assessed by Visual Analogue Scale (VAS)
Description: as for outcome 2
Time Frame: 30 minutes after regional anesthesia
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 15 | 28
units on a scale | 2.37 (2.33) | 1.77 (2.05)

5. Secondary Outcome: Success of Analgesia as Indicated by Pain Score Assessed by Visual Analogue Scale (VAS)
Description: as for outcome 2
Time Frame: 60 minutes after regional anesthesia
Population: Data for 1 participant in the epidural arm were not recorded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 14 | 28
units on a scale | 1.79 (2.22) | 1.63 (2.15)

6. Secondary Outcome: Success of Analgesia as Indicated by Pain Score Assessed by Visual Analogue Scale (VAS)
Description: as for outcome 2
Time Frame: 24 hours after regional anesthesia
Population: Data for 3 participants in the epidural arm and 8 participants in the CSE arm were not recorded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 12 | 20
units on a scale | 3.5 (2.65) | 2.53 (2.58)

7. Secondary Outcome: Childbirth Experience as Assessed by a Visual Analogue Scale (VAS)
Description: Childbirth experience was assessed by a visual analogue scale (VAS) with a scale of 1 to 10, with higher scores indicating a better childbirth experience.
Time Frame: 24 hours after regional anesthesia
Population: Data for 3 participants in the epidural arm and 8 participants in the CSE arm were not recorded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 12 | 20
units on a scale | 8.25 (2.63) | 9.25 (1.21)

8. Secondary Outcome: Maternal Satisfaction as Assessed by a Visual Analogue Scale (VAS)
Description: Maternal Satisfaction was assessed by a visual analogue scale (VAS) with a scale of 1 to 10, with higher scores indicating a higher level of satisfaction.
Time Frame: 24 hours after regional anesthesia
Population: Data for 3 participants in the epidural arm and 8 participants in the CSE arm were not recorded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 12 | 20
units on a scale | 8.42 (2.28) | 9.25 (1.59)

9. Secondary Outcome: Neonatal Outcome as Assessed by (APGAR) Score
Description: Apgar score is a method to quickly summarize the health of newborn children. The Apgar scale is determined by evaluating the newborn baby on five simple criteria [Appearance (skin color), Pulse (heart rate), Grimace (reflex irritability), Activity (muscle tone), and Respiration]. Each crtieria is rated on a scale from 0 to 2, then summing up the five values thus obtained. The resulting Apgar total score ranges from zero to 10. Scores of 7 and above are generally normal, 4 to 6 fairly low, and 3 and below are generally regarded as critically low.
Time Frame: 1 minute after birth
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 15 | 28
units on a scale | 8.60 (0.51) | 8.39 (0.69)

10. Secondary Outcome: Neonatal Outcome as Assessed by (APGAR) Score
Description: as for outcome 9
Time Frame: 5 minutes after birth
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 15 | 28
units on a scale | 8.93 (0.26) | 9.04 (0.19)

11. Secondary Outcome: Time From Regional Anesthesia to Delivery
Time Frame: from regional anesthesia to delivery (about 86 - 1205 minutes)
Population: For 2 participants in the CSE group, delivery time was not recorded and so the time from regional anesthesia to delivery could not be determined.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 15 | 26
minutes | 415.7 (208.2) | 454.5 (279.1)

12. Secondary Outcome: Time From Second Stage of Labor to Delivery
Description: The second stage of delivery begins after the cervix has dilated to 10 centimeters (cm).
Time Frame: from the second stage of labor to delivery (about 6 to 174 minutes)
Population: Because 2 in the epidural arm and 6 in the CSE arm never dilated to 10cms and were c-sectioned, it was not possible to obtain this value for these 8 participants. For 1 in the epidural arm and 1 in the CSE arm, delivery time was not recorded and so the time from the second stage of labor to delivery could not be determined for these 2 participants.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
Number analyzed (Participants) | 12 | 21
minutes | 71.25 (49.93) | 42.57 (44.82)

ADVERSE EVENTS:
Time Frame: 24 hours after regional anesthesia
Arm/Group | Epidural Anesthesia | Combined Spinal and Epidural (CSE) Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/28
Other Adverse Events (participants affected / at risk) | 5/15 | 4/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural Anesthesia (N=15) | Combined Spinal and Epidural (CSE) Anesthesia (N=28)
hypotension (Cardiac disorders) | 1 (1) | 1 (1)
nausea (General disorders) | 3 (3) | 1 (1)
vomiting (General disorders) | 1 (1) | 1 (1)
headache (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
lower than expected sample size (the study was powered for 60 but only 46 participants were enrolled)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT02105558/Prot_SAP_000.pdf